CLINICAL TRIAL: NCT06766214
Title: Augmentation Von Online-Psychotherapie Mit tDCS Bei Der Aufmerksamkeitsdefizit-/Hyperaktivitätsstörung (ADHS)
Brief Title: Attexis and tDCS for the Treatment of ADHD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Collaborators: Sooma Medical (Unknown); Gaia AG (Industry)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., Clinical Professor, MD, PhD, University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-3862-101
Record Dates: First submitted 2024-11-22; First posted 2025-01-09 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: ADHD
Keywords: ADHD; tDCS; Attexis; Psychotherapy; Home-based
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: 1. treatment with Attexis and tDCS and 2. treatment with Attexis and placebo tDCS
Who Masked: Investigator
Masking Description: https://www.random.org/lists/
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attexis and tDCS (Experimental): 15 patients receive three-month access to the psychotherapy app attexis and a tDCS device from the company Sooma, which is set to verum
  Interventions: Device: transcranial direct current stimulation
- Attexis and placebo-tDCS (Placebo Comparator): 15 patients receive three-month access to the psychotherapy app attexis and a tDCS device from the company Sooma, which is set to sham
  Interventions: Device: sham transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Simultaneous treatment with tDCS and online-based psychotherapy
  Other Names: attexis
  Arms: Attexis and tDCS
Device: sham transcranial direct current stimulation — Simultaneous treatment with sham-tDCS and online-based psychotherapy
  Other Names: attexis
  Arms: Attexis and placebo-tDCS

SUMMARY:
A randomized controlled two-arm study (RCT) will be conducted. It is planned to randomly assign eligible patients who receive a three-month access to the psychotherapeutic program (Attexis) to either an additional verum-tDCS or placebo-tDCS condition.

DETAILED DESCRIPTION:
The aim of this study is to determine whether the effectiveness of the home-based therapy program "Attexis" can be augmented with another home-based procedure, tDCS treatment, in order to achieve even higher improvement rates in the treatment of ADHD in the future. Before the actual start of treatment with Attexis, the presence of an ADHD diagnosis (ICD-10: F90.0) is checked by qualified medical staff at Medbo Regensburg. If the screened patient then meets the other inclusion criteria for Attexis and tDCS, he or she will be randomly assigned to either the intervention group (receives access to both Attexis and tDCS) or the placebo group (receives access to both Attexis and placebo tDCS). Based on the study by Schlechter et al. (2023), it is planned to treat patients receiving (placebo) tDCS treatment with 60 sessions (2mA, 20 minutes per day) by stimulating the left DLPFC. As patients will have a three-month access to Attexis, it is planned to administer the additional (placebo) tDCS treatment at the same time. As soon as a patient registers for the study, the safety aspects and inclusion/exclusion criteria for tDCS treatment are also checked in an initial interview after the ADHD diagnosis has been verified. The patient is then randomly assigned to one of the two study arms. A suitable appointment is then arranged for the patient to be admitted to the device. About 60 minutes are scheduled for the explanation and instruction of the tDCS device. During the appointment, an initial trial treatment is carried out so that the patient can get used to the treatment. All subsequent home-based treatments are carried out from Monday to Friday (each lasting 20 minutes) with video observation during the first week of treatment. For the sessions via teletherapy, software approved for clinical use (CLICKDOC version 5.9.1, La-Well Systems GmbH, CompuGroup Medical SE & Co. KGaA, Bünde, Germany) is to be used. At the end of the tDCS treatment, a final consultation will be arranged, which will take about 45 minutes. A follow-up (clinical ratings and attention test) will be carried out after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Gender: female, male, non-binary
* Age: 18 - 65
* Diagnosis of ADHD according to ICD-10
* ADHD severity score (cut-off): Score of ≥17 on either the inattention subscale or the impulsivity/hyperactivity subscale of the ASRS v1.1
* Stable treatment (psychotherapy, medication, no treatment, ...) (if applicable) for at least 30 days at the time of admission
* Consent to participate
* Sufficient knowledge of the German language

Exclusion Criteria:

tDCS:

* Fulfillment of the contraindications for tDCS (electrical implants or metallic objects in the body such as pacemakers or insulin pumps, skin diseases on the head)
* Neurological diseases (e.g. cerebrovascular events, neurodegenerative diseases, epilepsy, brain malformation, history of severe head injuries)
* Participation in another study during treatment
* Pregnancy or breastfeeding

Attexis:

* Diagnosis of a comorbid clinically relevant severe psychiatric disorder (severe affective disorder, autism spectrum disorder, psychotic disorder, borderline personality disorder, antisocial personality disorder, substance use disorder, suicidality)
* Plan to change an ongoing treatment (psychotherapy, medication, ...) in the next three months after enrollment in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Compliance (Number of days (60) of actual (Placebo-)tDCS-treatment) | 12 weeks
  Number of days of treatment with (Placebo-)tDCS
Efficacy 1 (Number of responders according to the ASRS-v1.1) | 12 weeks
  (Number of responders according to the ASRS-v1.1)
Efficacy 2 (Number of responders according to the subscale attention of the ASRS-v1.1) | 12 weeks
  Number of responders according to the subscale attention of the ASRS-v1.1
Efficacy 3 (Number of responders according to the subscale hyperactivity of the ASRS-v1.1) | 12 weeks
  Number of responders according to the subscale hyperactivity of the ASRS-v1.1
Stability of effects (Number of responders according to the change of the final ASRS-v1.1 sumscore) | 24 weeks
  Number of responders according to the change of the ASRS-v1.1 sumscore after treatment

SECONDARY OUTCOMES:
Adult ADHD Self-Report Scale Symptom Checklist (ASRS-v1.1, sumscore) | 12 weeks
  Adult ADHD Self-Report Scale Symptom Checklist (ASRS-v1.1) (the less the better) (sumscore: 0-72)
Adult ADHD Self-Report Scale Symptom Checklist (ASRS-v1.1, Subscale: Attention) | 12 weeks
  Adult ADHD Self-Report Scale Symptom Checklist (ASRS-v1.1) (the less the better) (subscale A: 0-36)
Adult ADHD Self-Report Scale Symptom Checklist (ASRS-v1.1, Subscale: hyperactivity) | 12 weeks
  Adult ADHD Self-Report Scale Symptom Checklist (ASRS-v1.1) (the less the better) (subscale B: 0-36)
Usability (sumscore of the Usability experience questionnaire UEQ) | 12 weeks
  Sumscore of the usability experience questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, PhD, Principal Investigator — University of Regensburg
Locations (1):
- Department of Psychiatry and Psychotherapy, University of Regensburg, Regensburg, Germany, Regensburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided